CLINICAL TRIAL: NCT07403526
Title: Transforming Global Surgery Capacity and Capability Through Affordable Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-102
Record Dates: First submitted 2025-02-20; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Hysterectomy (MeSH nr: E04.950.300.399)
Keywords: Virtual Reality; Simulation Training; Surgical Education; Postpartum Hemorrhage; Hysterectomy; Obstetric Surgical Procedures; Maternal Health Services; Global Health; Clinical Competence; Medical Education; Randomized Controlled Trial; Capacity Building; Educational Technology; Computer-Assisted Instruction; Skill Acquisition; Sub-Saharan Africa; Zambia; Low-Resource Settings
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) with a crossover design assessed the effectiveness of Deliberate VR Training for postpartum hysterectomy training.
  The intervention included a 9-day, structured VR-based training program, real-time feedback, and skill assessment. Surgical skill assessments were conducted using Objective Structured Assessment of Technical Skills (OSATS) scores, based on video recordings of surgical procedures on lifelike mannequins.
Who Masked: Outcomes Assessor
Masking Description: Evaluators assessing surgical performance using OSATS scores were blinded to group assignment to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deliberate Virtual Reality (VR) Training (Experimental): Participants in this arm underwent Deliberate Virtual Reality (VR) Training, a structured 9-day VR-based curriculum designed to improve surgical knowledge, technical skills, and confidence in performing postpartum hysterectomy. The training used interactive VR simulations, real-time performance feedback, and deliberate practice principles to enhance competency.
  Interventions: Behavioral: Deliberate Virtual Reality (VR) Training
- Standard Clinical Training (Active Comparator): Participants initially received standard clinical education on postpartum hysterectomy through traditional clinical training at their assigned hospitals. This included observation, supervised hands-on practice, and self-directed study without VR simulation. After completing the initial training phase, these participants crossed over to the Deliberate VR Training for an additional 9-day VR-based training program.
  Interventions: Behavioral: Standard Clinical Training

INTERVENTIONS:
Behavioral: Deliberate Virtual Reality (VR) Training — Deliberate VR Training is a self-guided, interactive virtual reality-based training program focused on surgical skill acquisition. The VR simulation includes step-by-step procedural guidance, performance tracking, and self-reflection exercises for postpartum hysterectomy training. Participants practiced daily, receiving objective feedback on surgical accuracy and technique. The intervention lasted 9 days, with 6-hour daily training sessions.
  Arms: Deliberate Virtual Reality (VR) Training
Behavioral: Standard Clinical Training — Standard Clinical Training followed a traditional mentor-based surgical training model at tertiary hospitals. Training included clinical observation, procedural discussions, and hands-on practice under supervision. Unlike the Deliberate VR group, participants did not have access to structured virtual reality simulation during the initial phase. Following post-training assessment, all participants in this arm crossed over to complete the Deliberate VR Training program.
  ________________________________________
  Arms: Standard Clinical Training

SUMMARY:
The goal of this randomized controlled trial was to evaluate whether Deliberate Virtual Reality (VR) training can improve surgical skills, knowledge, and confidence in performing postpartum hysterectomy among junior-level Zambian physicians in training.

The main questions it aims to answer are:

1. Can VR-based surgical training improve technical surgical skills in a real-world setting?
2. Does Deliberate VR training enhance knowledge retention and confidence compared to standard clinical training?

Study Design: Researchers randomly assigned participants to either:

1 Deliberate VR Training (intervention group): A 9-day VR-based surgical training program 2. Standard Training (control group): Conventional clinical education

Participants underwent assessments of surgical skills, knowledge, and confidence before and after training using objective structured assessment of technical skills (OSATS) and knowledge exams.

Key Findings:

1. The Deliberate VR group demonstrated significantly greater improvements in surgical knowledge, confidence, and OSATS scores compared to the standard training group.
2. VR training showed strong skill transfer to real-world surgical performance, suggesting that affordable and scalable VR training can help bridge surgical workforce gaps in resource-constrained settings.

This study highlights VR-based training as a potential scalable solution to strengthen surgical capacity in maternal health, addressing workforce shortages and improving equitable access to essential surgical care.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of Deliberate Virtual Reality (VR) Training as an innovative educational intervention for enhancing surgical skills, knowledge retention, and confidence in postpartum hysterectomy management among junior physicians in Zambia. The study employs a randomized controlled trial (RCT) with a crossover design, ensuring that all participants ultimately experience the VR training.

Study Rationale and Background: Postpartum hemorrhage (PPH) remains a leading cause of maternal mortality, particularly in low-resource settings where access to highly trained surgeons is limited. Traditional surgical training models rely on mentorship and hands-on experience, which may not be feasible in under-resourced clinical environments with limited faculty. Virtual reality offers a scalable, cost-effective alternative, allowing trainees to repeatedly practice surgical techniques in a controlled environment before real-world application.

Intervention Details: The Deliberate VR training model is a 9-day self-guided, simulation-based program designed to: Provide a structured, step-by-step approach to learning postpartum hysterectomy procedures. Utilize interactive VR environments that allow real-time assessment and feedback. Offer progress tracking and individualized goal-setting for surgical skill mastery. Incorporate reflection exercises to reinforce deliberate practice techniques.

Study Procedures: Participants were randomly assigned to two groups:

1. Intervention Group: Immediate Deliberate VR Training.
2. Control Group: Standard clinical training, followed by cross-over to VR training.

Outcomes:

1. Primary outcomes include surgical proficiency (measured via OSATS scoring) and knowledge acquisition.
2. Secondary outcomes assess confidence, skill retention, and real-world application in surgical settings.

Ethical Considerations: Ethical approval was obtained from University of Zambia Biomedical Research Ethics Committee, Southern Methodist University, University of North Carolina at Chapel Hill, and King's College London. Written informed consent was obtained from all participants. The study followed the Declaration of Helsinki guidelines for ethical research involving human participants.

Potential Impact The findings from this study may inform global health education strategies by demonstrating how low-cost VR interventions can strengthen surgical training, particularly in regions with surgical workforce shortages. If successful, this model could be adapted for other critical procedures and integrated into postgraduate medical training programs in resource-constrained settings.

ELIGIBILITY:
Inclusion Criteria:Participants were eligible for the study if they met the following criteria:

1. Junior-level Zambian physicians.
2. Recent graduates of the General Medical Officers (GMO) training program or first-year Obstetrics and Gynecology residents.
3. Within the first 18 months of their training at public hospitals in Lusaka, Zambia.
4. Actively involved in the clinical and surgical management of postpartum hemorrhage (PPH).
5. Available for the full duration of the 9-day training period.
6. Provided verbal agreement to participate after being informed about the study objectives and procedures.

Exclusion Criteria:

1. Previously completed formal postpartum hysterectomy training.
2. Had prior experience with virtual reality (VR)-based surgical training.
3. Unable to commit to the full 9-day training schedule.
4. Did not receive permission from clinical supervisors to participate.
5. Had a medical condition or visual impairment that prevented the use of VR equipment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Postpartum Hysterectomy Surgical Skill Performance | Baseline (pre-training) and post-training (Day 10)
  The primary outcome measure is the change in surgical skill performance as measured by Objective Structured Assessment of Technical Skills scale, a validated tool for assessing surgical performance. Scores are based on technical proficiency, respect for tissue, instrument handling, and procedural knowledge, as assessed by blinded evaluators reviewing video-recorded surgical performances on a high-fidelity mannequin. The Objective Structured Assessment of Technical Skills scale consists of seven subscales assessing different aspects of surgical performance. Each subscale is rated on a 5-point Likert scale (1 = poor performance, 5 = excellent performance). The total score is the sum of all seven subscales, ranging from 7 (lowest possible) to 35 (highest possible). Higher scores indicate better surgical skill performance.

SECONDARY OUTCOMES:
Change in Postpartum Hemorrhage Knowledge | Baseline and post-training (Day 10)
  Knowledge of postpartum hemorrhage management and postpartum hysterectomy procedures will be assessed using a 24-item multiple-choice Postpartum Hemorrhage Knowledge scale, developed from validated clinical content. Each question was either correct (1), or incorrect (0), with total scores ranging from 0 (low knowledge) to 24 (high knowledge).
Change in Surgical Confidence Ratings | Baseline and post-training (Day 10)
  Self-reported confidence in performing a postpartum hysterectomy, assessed using a 10-point Likert scale on three sub-scales measuring perceived (1) ability in surgical execution, (2) clinical decision-making, and (3) anatomical knowledge. Scores on each sub-scale ranged from 1 (very low confidence) to 10 (very high confidence).

OTHER OUTCOMES:
Correlation Between VR Training Engagement and Surgical Performance | Throughout the 9-day training period
  The correlation between time spent in VR training, number of simulation repetitions, and OSATS improvement will be analyzed to determine whether increased VR engagement leads to greater skill acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sullivan, MD, PhD, Principal Investigator — King's College London
Locations (1):
- University Teaching Hospital, Lusaka, Zambia, Zambia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to small sample size and participant confidentiality. The data collected includes sensitive training performance assessments and recorded surgical evaluations, which are not designed for public release.